CLINICAL TRIAL: NCT02534259
Title: Mobile Monitoring of Fracture Healing
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Gregory S. Lewis, Assistant Professor, Milton S. Hershey Medical Center
Other Study IDs: STUDY00002137
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Tibial Fractures
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Other: Force monitoring of external fixator struts

SUMMARY:
The objective of this study is to develop methods for using forces measured on circular external fixators to predict the state of individual patient's healing of severe tibial fractures and defects.

DETAILED DESCRIPTION:
Patients receiving external fixators for tibial fractures and defects will be recruited. Normal struts on the device will be substituted with similar but instrumented struts which enable force measurement. During clinical visits, forces in the fixator, plus foot forces, will be measured during ambulation. Changes in force measurements across treatment and bone healing will be analyzed.

Severe fractures in the lower limb are associated with high energy trauma in both civilian and military patients,and are sometimes treated with external fixation devices to stabilize the bone until healing has occurred. The devices are kept on the patient for up to a year or more at significant cost, intrusiveness, and risk of infection. The clinician must decide when to remove the device such that adequate healing has occurred and the bone will not re-fracture, but healing rates are variable and x-rays can be misleading. The clinician must also identify when a patient is starting to progress poorly and an early revision surgery is needed to prevent further complications.

The investigators' goal is to develop novel approaches for instrumenting and collecting mechanical data from orthopaedic braces and devices, and identifying new methodologies for interpreting this large volume of functional data for optimizing personalized treatment. The present study is focused on external fixators. Strain gauges will be adhered to the fixators so that fixator forces can be measured during clinical visits. In this pilot study the investigators will develop methods to predict healing based on these measured forces.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age
2. Patients scheduled to undergo or currently undergoing treatment at Hershey Medical Center for tibia fracture and/or defect using a circular external fixator including Ilizarov and Taylor Spatial Frame types.
3. Ability to perform study procedures including ambulation (with assistance device if needed)

Exclusion Criteria:

1. External fixator design that cannot be suitably instrumented for force measurements due to space constraints or other issues
2. Axially stable fracture
3. Inability to understand English
4. Inability to provide informed consent
5. Difficulty maintaining follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing treatment for severe tibia fracture and/or defect using a circular external fixator.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-08; Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Forces measured in the external fixator during ambulation during clinical visits | Approximately 5 times across treatment, with treatment lasting months to a year or more

SECONDARY OUTCOMES:
Forces measured in instrumented insoles during ambulation during clinical visits | Approximately 5 times across treatment, with treatment lasting months to a year or more
  Simultaneously measured during outcome 1 measurements

OTHER OUTCOMES:
Radiographic and other clinical assessment of bone healing during clinical visits | Approximately 5 times across treatment, with treatment lasting months to a year or more
  Simultaneously measured during outcome 1 measurements

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Lewis, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States